CLINICAL TRIAL: NCT04071054
Title: Optimized Continuous 7-day Detection of Arrhythmias in Dialysis Population by a Patch With a High Resolution Differentiation of Atrial Activity
Brief Title: Continuous 7-day Detection of Arrhythmias in Dialysis Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Guerkan SENGOELGE, Optimized continuous 7-day detection of arrhythmias in dialysis population by a patch with a high resolution differentiation of atrial activity, Medical University of Vienna
Other Study IDs: Continuous 7-day ECG
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Arrythmia; Dialysis; Complications
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis patients
  Interventions: Diagnostic Test: Carnation Ambulatory Monitor (CAM)

INTERVENTIONS:
Diagnostic Test: Carnation Ambulatory Monitor (CAM) — 7-day detection of arrhythmias with Carnation Ambulatory Monitor (CAM)

SUMMARY:
The Carnation Ambulatory Monitor (CAM) is an innovative diagnostic patch device that allows to differentiate the different kinds of arrhythmias more precisely than any other ECG-monitoring device. It attaches on the sternum and can be carried for a week without any breaks. This allows a continuous rhythm monitoring without any gap for 7 days.

This device will be used in dialysis patients to monitor arrhythmias during changes in volume and/or electrolyte balance due to dialysis, in the phases after dialysis as well as before dialysis in the short or long intervals between dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years.
* Written informed consent

Exclusion Criteria:

* Participation in another study within 4 weeks before study begin
* Pacemaker
* ICD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with a chronic hemodialysis program
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of dialysis patients with an arrhythmia | ECG monitoring over 7 days (3 intermittent hemodialysis sessions)
  Detection of arrhythmias (including distribution of ventricular and atrial arrhythmias) by means of Carnation Ambulatory Monitor (CAM) in hemodialysis patients during an entire week, thus including all different phases: during/after/before dialysis sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Vienna, Austria